CLINICAL TRIAL: NCT07050849
Title: The Effects of Slackline Training On Core Stabilization, Physical Performance and Balance In Young Adults
Brief Title: Effects of Slackline Training on Core Strength and Balance in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BÜŞRA ŞAHİN (Other)
Responsible Party: Sponsor-Investigator, BÜŞRA ŞAHİN, Research Assistant, Uludag University
Organization: Uludag University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-4/16
Record Dates: First submitted 2025-05-30; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Core Stability
Keywords: Core Stability; young adults; physical performance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slackliner Group (Experimental): Participants in this group received supervised slackline training sessions three times per week for six weeks. Each session lasted 45 minutes and included dynamic balance and core stabilization exercises performed on a slackline. A total of 18 sessions were conducted. The training was delivered by qualified instructors in a controlled indoor environment.
  Interventions: Behavioral: Slackline Training
- Control Group (No Intervention): Participants in this group did not receive any structured intervention during the study period. They were instructed to maintain their usual daily routines without engaging in any specific balance or core training activities. No supervised sessions or exercise protocols were applied.

INTERVENTIONS:
Behavioral: Slackline Training — This intervention consisted of a six-week supervised slackline training program designed to improve core stability, physical performance, and dynamic balance. Participants in the intervention group performed 18 sessions (3 sessions per week, 45 minutes each) using a Gibbon-brand slackline (12.5 meters in length, 50 mm wide). The training protocol included a structured progression of 11 exercises, ranging from assisted standing to unassisted long walks and dynamic movements on the slackline. All sessions were conducted under the supervision of a licensed physiotherapist to ensure participant safety and training fidelity. Exercises were adapted weekly to increase difficulty, challenge motor control, and stimulate neuromuscular adaptation.
  Arms: Slackliner Group

SUMMARY:
This study aims to examine the effects of slackline training on core strength, physical performance, and balance in healthy young adults. A total of 40 participants were randomly assigned to either a slackline training group or a control group. The training group completed supervised slackline sessions three times per week for six weeks. Various physical and balance tests were performed before and after the intervention. The results showed that slackline training improved core stability, physical performance, and dynamic balance. These findings suggest that slackline exercises may be a useful method to enhance physical function in young adults.

ELIGIBILITY:
Inclusion Criteria:

* University student status

Age between 18 and 27 years

Voluntary participation with signed informed consent

Physically healthy and able to participate in physical activities

Exclusion Criteria:

* Being a licensed or professional athlete

History of orthopedic injuries or surgery

Neurological or vestibular disorders affecting balance

Cardiovascular disease

Color blindness or visual impairments interfering with performance

Inability to participate in physical testing or training

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Core Stabilization Performance | Baseline to 6 weeks post-intervention
  Trunk Flexion Test: The participant was positioned with back support, knees and hips flexed at 90°, feet fixed on the bed, and arms crossed over the chest. The trunk was set at a 60° flexion angle from the bed. Before removing the back support, the participant was instructed to maintain the trunk position for as long as possible Trunk Extension Test: The participant was positioned with their spina iliaca anterior superior aligned with the edge of the bed. They were instructed to place their hands on opposite shoulders and maintain the upper trunk in a horizontal position for as long as possible Prone Bridge Test: The participant was positioned prone, with hands, elbows, and feet shoulder-width apart. They were then instructed to lift their pelvis off the bed and maintain this position using only the toes, forearms, and elbows as the support surfaces Side Bridge Test: The participant was positioned on their dominant side on the bed, with the support arm flexed at the elbow, knees and

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The decision regarding IPD sharing has not yet been made. The availability of de-identified data will depend on institutional policies, ethical considerations, and potential requests after publication.

REFERENCES:
- [Background] Donath L, Roth R, Zahner L, Faude O. Slackline Training (Balancing Over Narrow Nylon Ribbons) and Balance Performance: A Meta-Analytical Review. Sports Med. 2017 Jun;47(6):1075-1086. doi: 10.1007/s40279-016-0631-9. PMID 27704483